CLINICAL TRIAL: NCT02815800
Title: Efficacy of Ethnodyne Visio in Parkinson's Disease
Acronym: ETHNOPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: ETHNODYNE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6312
Record Dates: First submitted 2016-06-13; First posted 2016-06-28 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Parkinson's Disease
Keywords: Treatment; Motor signs; Non motor signs; Fluctuations; Open labelled
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ETHNODYNE VISIO (Experimental): Administration 2 times a day of a dietary supplement, as add on therapy, in patients with Parkinson s disease
  Interventions: Dietary Supplement: ETHNODYNE VISIO

INTERVENTIONS:
Dietary Supplement: ETHNODYNE VISIO

SUMMARY:
ETHNODYNE VISIO is a food supplement composed of an innovative plant-based active ingredient acting alongside vitamin B2. It is proposed in patients with visual problems. Based on clinical and experimental data, the investigators propose a pilot open study in order to test the efficacy of "Ethnodyne visio" in patients with Parkinson 's disease (PD). The hypothesis is that Ethnodyne visio may improve motor and non motor signs of PD. 24 patients with PD will be evaluated before and after 3 months of add on treatment by Ethnodyne visio.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson disease (PD) with at least 3 years of evolution
* Hoehn and Yahr score 2 or 3
* with moderate fluctuations (score 1 or 2 for item 3 score IV MSD UPDRS)
* with no modification in anti-parkinsonian drugs since at least 1 month
* minimental test >24

Exclusion Criteria:

* known intolerance to Ethnodyne visio
* woman of childbearing potential or breastfeeding
* anticipated anti-parkinsonian treatment modification during the 3 months of the study
* antidepressant or anxiolytic drugs modified within one month prior to inclusion visit
* other chronic disease
* concomitant participation in a another clinical trial
* Subject under legal guardianship

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Change in MDS UPDRS III score | baseline and following 3 months of treatment

SECONDARY OUTCOMES:
Change in MDS UPDRS I, II and IV score | baseline and following 3 months of treatment
Change in Levodopa equivalent dose treatment (equivalence table) | baseline and following 3 months of treatment
Frequency, seriousness and severity of adverse event reactions | during the 3 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurologie,Hôpital de Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No